CLINICAL TRIAL: NCT06720688
Title: Association Between Ultrasound Morphology of Intestinal Endometriosis Nodules and Symptom Severity
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOSIGNS
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis Rectum
Keywords: Endometriosis; Ultrasound; Gynaecology
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Association between the ultrasound appearance of deep bowel endometriosis and the frequency of pain

DETAILED DESCRIPTION:
In order to improve the diagnostic power of the ultrasound method, it is important to evaluate the association between the ultrasound appearance of the nodule of intestinal deep endometriosis and the frequency of pain, thus assessing the prevalence of moderate or severe clinical symptoms, in patients with newly diagnosed intestinal deep endometriosis, according to the ultrasound morphology of the posterior deep endometriosis nodule proposed in the International Deep Endometriosis Analysis Group (IDEA) Consesus.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years;
* Presence of posterior rectus intestinal deep endometriosis confirmed on TV ultrasound between 01/01/2018 and 30/06/2023;
* Informed consent obtained

Exclusion Criteria:

* Virgo patients;
* Patients reporting intolerance to transvaginal ultrasound;
* Current or history of gynaecological oncology;
* Previous surgery of the sigma and rectum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an ultrasound diagnosis of deep bowel endometriosis undergoing surgery and patients who are not candidates for surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of moderate or severe clinical symptoms | At diagnosis or in the previous 6 months
  Prevalence of moderate or severe clinical symptoms in patients with newly diagnosed deep bowel endometriosis according to the ultrasound morphology of the posterior deep endometriosis nodule proposed in the IDEA Consensus.

SECONDARY OUTCOMES:
Ultrasound morphologies of the intestinal endometriosis nodule and the frequency of associated lesions | At diagnosis or in the previous 6 months
  Calculate the proportion of ultrasound morphologies of the intestinal endometriosis nodule and the frequency of associated lesions (adenomyosis, anterior endometriosis, parametrial, LUS).
Association between ultrasound morphology and specific clinical symptoms | At diagnosis or in the previous 6 months
  Check whether the different categories of ultrasound morphology, described in the IDEA Consensus, are associated with specific clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Diego Raimondo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy